CLINICAL TRIAL: NCT05968482
Title: A Phase 1, Single-Center, Randomized, Open-Label, Bioavailability and Safety Three Period Crossover Multiple-Dose Study Comparing Two Dose Levels of AMZ001 (Diclofenac Sodium Gel 3.06%) and One Dose Level of Diclofenac Sodium 1% Gel in Healthy Subjects
Brief Title: Bioavailability and Safety Study Comparing Two Dose Levels of AMZ001 and One Dose Level of Diclofenac Sodium 1% Gel in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amzell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMZ001-008
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AMZ001 Low dose (Experimental): AMZ001 applied once daily for 7 consecutive days
  Interventions: Drug: Diclofenac Sodium Gel
- AMZ001 High dose (Experimental): AMZ001 applied once daily for 7 consecutive days
  Interventions: Drug: Diclofenac Sodium Gel
- Diclofenac Sodium 1% Gel (Active Comparator): Reference product applied four-times daily for 7 consecutive days
  Interventions: Drug: Diclofenac Sodium Gel

INTERVENTIONS:
Drug: Diclofenac Sodium Gel — Topical application on both knees

SUMMARY:
The goal of this clinical trial is to compare drug exposure from two different products (AMZ001 and Diclofenac Sodium 1% Gel) in healthy participants on Day 7 after repeated topical administrations for 7 days.

Participants will receive, in a crossover design, three different treatments

* AMZ001 Low dose
* AMZ001 High dose
* Diclofenac Sodium 1% Gel

Safety and tolerability of AMZ001 will be also investigated.

DETAILED DESCRIPTION:
On their both knees, participants will apply once daily either low dose of AMZ001 or high dose of AMZ001 for 7 consecutive days. Participants will also apply Diclofenac Sodium 1% Gel as per label information on each knee.

Intensive pharmacokinetic assessment (blood samplings) will be performed on the first day of application (Day 1) as well as on the last day of application (Day 7).

Each participant will receive each of the three treatments in a randomized manner. Between each treatment, participant will not receive any of the three tested therapies between 3 weeks before receiving the next therapy. (washout period)

Participants will stay on the clinical unit only during each period of treatment but not during washout period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants 18-65 years of age (e.g., in general good physical health, as judged by the Investigator and no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG (electrocardiogram) or clinical laboratory tests)
* Has a body mass index (BMI) between 18.0 and 35.0 kg/m^2 (kilogram per square meter) at Screening.
* In the case of females of child-bearing potential ([FCBP) unless surgically sterilized [hysterectomy, bilateral oophorectomy, bilateral tubal ligation] or are postmenopausal for at least 12 months), are using two acceptable forms of birth control (hormonal contraceptives i.e., oral/implant/injectable/transdermal; intrauterine device (IUD) and/or barrier methods [female condom, male condom, diaphragm, cervical cap, spermicide]; note: 2 barrier methods are two acceptable forms of birth control)). Abstinence or partner's vasectomies are acceptable if the female participant agrees to implement two acceptable forms of birth control if her lifestyle/partner changes.
* Females of child-bearing potential have a negative serum pregnancy test (SPT) at Screening and negative urine pregnancy test (UPT) on Day -1 of each period and at end of treatment (EOT) visit
* Are free of any systemic or dermatologic disorder and chronic or acute infections, which, in the opinion of the Principal Investigator (PI), will interfere with the study results or increase the risk of adverse events (AEs)
* Read, understand, and provide signed informed consent before any assessment is performed.

Exclusion Criteria:

* Participant has any visible skin disease, skin lesions, wounds, or a significant amount of hair at the application site (knee)
* Use of an investigational medicinal product (IMP) within 30 days or 5 half-lives (if known), whichever is longer, of enrollment or during the study.
* Treated with systemic or local diclofenac within 30 days of enrollment or during the study (except for study IMP)
* Known hypersensitivity to diclofenac, aspirin, Xarelto, coumadin, or other non-steroidal anti-inflammatory drugs (NSAIDs), including Cyclooxygenase-2 (COX-2) inhibitors.
* Any history of drug hypersensitivity, asthma, urticaria, or other significant allergic diathesis. Participants with uncomplicated seasonal allergic rhinitis can be accepted only if the expected allergy season is clearly outside enrollment / treatment periods.
* Females who are pregnant and/or lactating
* Of child-bearing potential but not willing to use adequate contraception for the duration of the study
* Participant is a current smoker and unable to abstain from smoking during the treatment periods.
* Use of any topical medication, cosmetics, cream, ointments, lotions on the treatment site 1 week prior to enrollment through EOT visit
* Use of any medication (including over-the-counter medication, dietary supplements, and herbal remedies) within 2 weeks before first scheduled study drug administration or within less than 5 times the elimination half-life of the respective drug (whichever is longer) or is anticipated to require concomitant medication during the 2-week period or at any time throughout the study. Consumption of any drug metabolizing enzyme (e.g., cytochrome P450 3A4 (CYP3A4) or other cytochrome P450 enzymes) inducing or inhibiting beverages or food (e.g., broccoli, Brussel sprouts, grapefruit, grapefruit juice, star fruit) within 3 days prior to and during each treatment period
* Participant has a known or suspected malignancy, excluding basal cell cancer unless it is associated with the treatment area.
* Participant has a positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C antibody (Anti-HCV)
* Participant has any acute or chronic condition or is using medications, which, in the investigator's opinion, would make it unsafe for the participant to participate in this study, including clinically significant abnormal laboratory values, vital signs, physical examination findings prior to randomization or during study participation.
* History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine (greater than (>) 1.43 mg/dL (milligram per deciliter)) or blood urea nitrogen (greater than or equal to (≥) 35 mg/dL) or the presence of clinical significant abnormal urinary constituents (e.g., albuminuria)
* History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A participant will be excluded if more than one of the following lab value deviations are found: 1) aspartate aminotransferase (AST) (≥ 1.5 upper limit of normal (ULN)), alanine aminotransferase (ALT) (≥ 1.5 ULN), 2) Gamma-Glutamyl Transferase (GGT) (≥ 1.5 ULN), alkaline phosphatase (ALP) (≥ 1.5 ULN), 3) total bilirubin (> 2.00 mg/dL) or creatine kinase (≥ 3 ULN). A single deviation from the above values is acceptable and will not exclude the participant, unless specifically advised by the Investigator.
* Participant has clinically relevant chronic or acute infectious illnesses or febrile infections within 2 weeks prior to the first scheduled study drug administration
* Participant has gastrointestinal bleeding issues, e.g., Gastroesophageal Reflux Disease (GERD), Peptic Ulcer Disease (PUD)
* Participant has a hospital admission or major surgery within 30 days prior to randomization.
* Participant has a donation or blood collection of more than 1 unit (approximately 450 mL(milliliter)) of blood (or blood products) or acute loss of blood during the 30 days prior to randomization.
* Participant has a history of alcohol abuse, prescription drug abuse, or illicit drug use within 6 months prior to Screening.
* Participant meets eligibility criteria, but study is filled
* Participant who is an investigational site staff member directly involved in the conduct of the study and his/her family members, site staff member otherwise supervised by the Investigator, or participant who is a Amzell B.V. employee directly involved in the conduct of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AMZ001 Low / AMZ001 High / Diclofenac: Participants first received AMZ001 Low dose applied once daily for 7 days (Period 1). After a washout period of at least 21 days, they then received AMZ001 high dose applied once daily for 7 days (Period 2). After another washout period of at least 21 days, they finally received Diclofenac Sodium 1% Gel applied four times daily for 7 days (Period 3). At the end of Period 3, there will be three additional PK blood samples taken respectively at 3 weeks (21 days), 4 weeks (28 days), and 5 weeks (35 days) after the last application to compare elimination phase of AMZ001 vs. Diclofenac Sodium 1% Gel
- Diclofenac/AMZ001 High/AMZ001 Low: Participants first received Diclofenac Sodium 1% Gel applied four times daily for 7 days. After a washout period of at least 21 days, they then received AMZ001 high dose applied once daily for 7 days. After another washout period of at least 21 days, they finally received AMZ001 Low dose applied once daily for 7 days. At the end of Period 3, there will be three additional PK blood samples taken respectively at 3 weeks (21 days), 4 weeks (28 days), and 5 weeks (35 days) after the last application to compare elimination phase of AMZ001 vs. Diclofenac Sodium 1% Gel
- Diclofenac/AMZ001 Low/AMZ001 High: Participants first received Diclofenac Sodium 1% Gel applied four times daily for 7 days. After a washout period of at least 21 days, they then received AMZ001 Low dose applied once daily for 7 days. After another washout period of at least 21 days, they finally received AMZ001 high dose applied once daily for 7 days. At the end of Period 3, there will be three additional PK blood samples taken respectively at 3 weeks (21 days), 4 weeks (28 days), and 5 weeks (35 days) after the last application to compare elimination phase of AMZ001 vs. Diclofenac Sodium 1% Gel
- AMZ001 High/AMZ001 Low/Diclofenac: Participants first received AMZ001 High dose applied once daily for 7 days. After a washout period of at least 21 days, they then received AMZ001 low dose applied once daily for 7 days. After another washout period of at least 21 days, they finally received Diclofenac Sodium 1% Gel applied four times daily for 7 days. At the end of Period 3, there will be three additional PK blood samples taken respectively at 3 weeks (21 days), 4 weeks (28 days), and 5 weeks (35 days) after the last application to compare elimination phase of AMZ001 vs. Diclofenac Sodium 1% Gel
- AMZ001 Low/Diclofenac/AMZ001 High: Participants first received AMZ001 low dose applied once daily for 7 days. After a washout period of at least 21 days, they then received Diclofenac Sodium 1% Gel applied four times daily for 7 days. After another washout period of at least 21 days, they finally received AMZ001 high dose applied once daily for 7 days. At the end of Period 3, there will be three additional PK blood samples taken respectively at 3 weeks (21 days), 4 weeks (28 days), and 5 weeks (35 days) after the last application to compare elimination phase of AMZ001 vs. Diclofenac Sodium 1% Gel
- AMZ001 High/Diclofenac/AMZ001 Low: Participants first received AMZ001 high dose applied once daily for 7 days. After a washout period of at least 21 days, they then received Diclofenac Sodium 1% Gel applied four times daily for 7 days. After another washout period of at least 21 days, they finally received AMZ001 low dose applied once daily for 7 days. At the end of Period 3, there will be three additional PK blood samples taken respectively at 3 weeks (21 days), 4 weeks (28 days), and 5 weeks (35 days) after the last application to compare elimination phase of AMZ001 vs. Diclofenac Sodium 1% Gel
Period: First Crossover Period
Arm/Group | AMZ001 Low / AMZ001 High / Diclofenac | Diclofenac/AMZ001 High/AMZ001 Low | Diclofenac/AMZ001 Low/AMZ001 High | AMZ001 High/AMZ001 Low/Diclofenac | AMZ001 Low/Diclofenac/AMZ001 High | AMZ001 High/Diclofenac/AMZ001 Low
Started | 12 | 12 | 12 | 13 | 13 | 12
Completed | 12 | 12 | 11 | 13 | 13 | 11
Not Completed | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Period: Second Crossover Period
Arm/Group | AMZ001 Low / AMZ001 High / Diclofenac | Diclofenac/AMZ001 High/AMZ001 Low | Diclofenac/AMZ001 Low/AMZ001 High | AMZ001 High/AMZ001 Low/Diclofenac | AMZ001 Low/Diclofenac/AMZ001 High | AMZ001 High/Diclofenac/AMZ001 Low
Started | 12 | 12 | 11 | 13 | 13 | 11
Completed | 12 | 12 | 11 | 13 | 12 | 11
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Third Crossover Period
Arm/Group | AMZ001 Low / AMZ001 High / Diclofenac | Diclofenac/AMZ001 High/AMZ001 Low | Diclofenac/AMZ001 Low/AMZ001 High | AMZ001 High/AMZ001 Low/Diclofenac | AMZ001 Low/Diclofenac/AMZ001 High | AMZ001 High/Diclofenac/AMZ001 Low
Started | 12 | 12 | 11 | 13 | 12 | 11
Completed | 12 | 11 | 11 | 13 | 11 | 11
Not Completed | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — failure to meet continuation criteria | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AMZ001 Low/AMZ001 High/Diclofenac: Low/High/Diclofenac
- Diclofenac/AMZ001 High/AMZ001 Low: Diclofenac/High/Low
- Diclofenac/AMZ001 Low/AMZ001 High: Diclofenac/Low/High
- AMZ001 High/AMZ001 Low/Diclofenac: High/Low/Diclofenac
- AMZ001 Low/Diclofenac/AMZ001 High: Low/Diclofenac/High
- AMZ001 High/Diclofenac/AMZ001 Low: High/Diclofenac/Low
- Total: Total of all reporting groups
Arm/Group | AMZ001 Low/AMZ001 High/Diclofenac | Diclofenac/AMZ001 High/AMZ001 Low | Diclofenac/AMZ001 Low/AMZ001 High | AMZ001 High/AMZ001 Low/Diclofenac | AMZ001 Low/Diclofenac/AMZ001 High | AMZ001 High/Diclofenac/AMZ001 Low | Total
Number analyzed (Participants) | 12 | 12 | 12 | 13 | 13 | 12 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (11.20) | 42.3 (14.69) | 36.4 (12.35) | 42.3 (10.60) | 39.8 (11.98) | 41.8 (13.47) | 41.1 (12.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 5 | 10 | 7 | 4 | 38
  Male | 5 | 7 | 7 | 3 | 6 | 8 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 5 | 8 | 4 | 4 | 27
  Not Hispanic or Latino | 9 | 9 | 7 | 5 | 9 | 8 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 0 | 1 | 3
  Black or African American | 6 | 6 | 7 | 5 | 6 | 7 | 37
  White | 5 | 6 | 4 | 7 | 7 | 3 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Compare Exposure to Diclofenac
Description: Area under the curve (AUC) from time zero to 24 hours
Time Frame: Day 7
Population: All subjects for which at least AUC0-τ or Cmax can be determined for the reference treatment (Diclofenac Sodium 1% Gel) along with at least one of Treatments AMZ001 Low dose or AMZ001 High dose are included in the analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- AMZ001 Low Dose: AMZ001 Low dose received either during Period 1, Period 2 or Period 3
- AMZ001 High Dose: AMZ001 High dose received either during Period 1, Period 2 or Period 3
- Diclofenac Sodium 1% Gel: Reference product applied four-times daily for 7 consecutive days received either in Period 1, Period 2 or Period 3
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
ng*hr/mL | 141.5 (89.8) | 166.1 (90.3) | 202.3 (79.4)

2. Primary Outcome: Pharmacokinetic Parameter - Cmax
Description: Maximum plasma drug concentration (Cmax)
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
ng/mL | 4.66 (122.4) | 6.22 (128.9) | 3.85 (122.2)

3. Secondary Outcome: Pharmacokinetic Parameter - Cmin
Description: Minimum plasma drug concentration (Cmin)
Time Frame: Day 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
ng/mL | 3.09 (96.3) | 3.38 (90.1) | 5.03 (80.1)

4. Secondary Outcome: Pharmacokinetic Parameter - Tmax
Description: Time to reach maximum plasma concentration (Tmax)
Time Frame: Day 7
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
hr | 8 [2 to 24] | 10 [2 to 24] | 18 [2 to 24]

5. Secondary Outcome: Pharmacokinetic Parameter - Ke
Description: Terminal disposition rate constant (Ke)
Time Frame: Day 7
Population: All subjects for which at least AUC0-τ or Cmax can be determined for the reference treatment (Diclofenac Sodium 1% Gel) along with at least one of Treatments AMZ001 Low dose or AMZ001 High dose are included in the analysis population.
  Analysis specified that Ke would be determined whenever the elimination phase after the Day 7 dose appeared to be adequately sampled based on a visual inspection of the log-linear plots.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
1/hr | NA (NA) — The PK parameter was not determined because high variability during the elimination phase did not permit linear regression analysis with sufficient confidence. inspection of the individual subject plots of diclofenac concentration vs time post-dose show that the curves are too variable to allow a linear regression analysis. | NA (NA) — The PK parameter was not determined because high variability during the elimination phase did not permit linear regression analysis with sufficient confidence. inspection of the individual subject plots of diclofenac concentration vs time post-dose show that the curves are too variable to allow a linear regression analysis. | NA (NA) — The PK parameter was not determined because high variability during the elimination phase did not permit linear regression analysis with sufficient confidence. inspection of the individual subject plots of diclofenac concentration vs time post-dose show that the curves are too variable to allow a linear regression analysis.

6. Secondary Outcome: Pharmacokinetic Parameter - Cavg
Description: Average plasma concentration (Cavg)
Time Frame: Day 7
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
ng/mL | 5.90 (89.8) | 6.92 (90.3) | 8.43 (79.4)

7. Secondary Outcome: Pharmacokinetic Parameter - Tmax
Description: Time to reach maximum plasma concentration
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
hr | 14 [2 to 24] | 16 [4 to 24] | 20 [6 to 24]

8. Secondary Outcome: Pharmacokinetic Parameter - Cavg
Description: Average plasma concentration (Cavg)
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 69 | 69 | 69
ng/mL | 2.59 (119.8) | 3.48 (124.8) | 1.60 (109.9)

9. Secondary Outcome: Local Tolerability
Description: Incidence of application site reactions according to the terminology of the International Contact Dermatitis Research Group
Time Frame: Day 1 to Day 7
Population: The Safety population includes randomized subjects who received at least one dose of AMZ001 Low dose or High dose or Diclofenac Sodium 1% Gel
Measure: Count of Participants; unit: Participants
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
Number analyzed (Participants) | 71 | 72 | 72
Participants
  no skin reaction | 62 | 61 | 64
  doubtful skin reaction | 7 | 7 | 7
  mild skin erythema | 1 | 4 | 1
  strong skin erythema | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From initiation of first period (Day 1) to completion of last period (Day 98)
Arm/Group | AMZ001 Low Dose | AMZ001 High Dose | Diclofenac Sodium 1% Gel
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 7/71 | 8/72 | 5/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMZ001 Low Dose (N=71) | AMZ001 High Dose (N=72) | Diclofenac Sodium 1% Gel (N=72)
Administration site dermatitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion / abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Administration site dryness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Administration site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site dermatitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 3 (3) | 1 (1)
Application site hypersensitivity (General disorders) | 0 (0) | 2 (2) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratinosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Master Service agreement: Work Product shall be and remain the sole and exclusive property of Sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT05968482/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT05968482/SAP_001.pdf